CLINICAL TRIAL: NCT06713057
Title: Precision Medicine Applied to Locally Advanced or Metastatic Poorly Differentiated or Anaplastic Thyroid Cancer Using Tumor Derived Organoids and In-vitro Sensitivity Testing: a Phase 2, Single-center, Open-label, and Non-comparative Study
Brief Title: Efficacy of Organoid-Based Chemotherapy Drug Precision Screening to Guide Treatment for Thyroid Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Li Zhihui, Dean of the Thyroid Surgery Department, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX20231471
Record Dates: First submitted 2024-11-25; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Locally Advanced Thyroid Gland Carcinoma; Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Vindesine; Cisplatin; Doxorubicin; Cyclophosphamide; Docetaxel; CP protocol; Paclitaxel; TP protocol; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Organoid-guided chemotherapeutic group (Experimental): Patients who take the recommended chemothetapy drugs regularly based on sensitivity analysis.
  Interventions: Drug: Cyclophosphamide+Pemetrexed+5-Fluorouracil; Drug: Cyclophosphamide+Doxorubicin+5-Fluorouracil; Drug: Vindesine + Cisplatin; Drug: Doxorubicin + Cisplatin; Drug: Doxorubicin + Cyclophosphamide + Cisplatin; Drug: Docetaxel + Doxorubicin; Drug: Paclitaxel + Carboplatin; Drug: Paclitaxel + Doxorubicin; Drug: Paclitaxel + Cisplatin; Drug: Gemcitabine alone

INTERVENTIONS:
Drug: Cyclophosphamide+Pemetrexed+5-Fluorouracil — IV or PO
Drug: Cyclophosphamide+Doxorubicin+5-Fluorouracil — IV or PO
Drug: Vindesine + Cisplatin — IV or PO
Drug: Doxorubicin + Cisplatin — IV or PO
Drug: Doxorubicin + Cyclophosphamide + Cisplatin — IV or PO
Drug: Docetaxel + Doxorubicin — IV or PO
Drug: Paclitaxel + Carboplatin — IV or PO
Drug: Paclitaxel + Doxorubicin — IV or PO
Drug: Paclitaxel + Cisplatin — IV or PO
Drug: Gemcitabine alone — IV or PO

SUMMARY:
The current study aims to explore the potential advantages of chemotherapy that is implemented based on drug sensitivity testing. This pertains to individuals with locally advanced or metastatic poorly differentiated or anaplastic thyroid cancer who have undergone conventional therapy in the past or unresectable patients .

DETAILED DESCRIPTION:
This research trial aims to determine the efficacy of organoid-guided chemotherapy for patients with locally advanced or metastatic poorly differentiated or anaplastic thyroid cancer.

Currently, there are numerous clinical trials evaluating various molecularly targeted therapies for refractory, poorly differentiated thyroid cancer. Preoperative personalized targeted neoadjuvant therapy has been established as a critical approach in managing advanced thyroid cancer. However, clinical trials investigating personalized chemotherapy to guide the treatment of thyroid cancer remain scarce.

Tumor organoids represent a sophisticated three-dimensional pathological model that preserves the histological and molecular characteristics of the original tumor. These models can be utilized to assess the in vitro efficacy of multiple anticancer drugs. The investigators' objective is to validate the effectiveness and safety of selecting and processing chemotherapeutic agents through drug susceptibility testing, thereby ensuring pragmatic and precise treatment tailored to individual patients' needs.

The investigators will also investigate the variables affecting the effectiveness of chemotherapy that is guided by organoids. Additionally, side effects related to the medication are also studied.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age on the day of signing informed consent
2. Cytologically confirmed thyroid neoplasm, including papillary thyroid carcinoma (PTC), follicular thyroid carcinoma (FTC), poorly differentiated thyroid carcinoma (PDTC), medullary thyroid carcinoma (MTC), anaplastic thyroid carcinoma (ATC)
3. Patients defined as poorly differentiated iodine-refractory thyroid tumors with inoperable locally advanced disease or metastases. The primary tumor may or may not be removed, but the risk of aerodigestive compression or bleeding should be excluded.
4. Evidence of extrathyroidal extension and/or locally invasive disease and deemed at risk for R2 resection by treating team on clinical and/or fiberoptic examination and/or radiographic evaluation in the primary or recurrent setting. Evidence of "at risk for R2 resection" includes:

   1. Vocal cord paralysis by fiberoptic examination
   2. Extrathyroid and/or extranodal extension on CT or MRI, including tracheal and/or laryngeal cartilage invasion, esophageal involvement, and/or involvement of perithyroid muscles (e.g. strap, sternocleidomastoid, inferior constrictor muscles) or bone involvement
   3. Extension into the mediastinum with visceral and/or vascular involvement
   4. Involvement of the carotid artery or other major vessel by 180 degrees or more (exclusive of complete encasement)
   5. Other factors that make the participant to be "at risk for R2 resection" may be allowed, after discussion with the study's principal investigator
5. At least one measurable lesion as defined by RECIST v1.1
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 and no medical contraindication to surgery
7. Surgical morbidity/complexity score of 1 to 4 (moderate, severe, very severe, or unresectable)
8. The expected survival time was more than 2 months
9. Adequate end-organ function (including bone marrow, coagulation, renal, liver and cardiac) 28 days prior to the study registration as defined below:

   1. leukocytes ≥3,000/mcL
   2. absolute neutrophil count ≥1,500/mcL
   3. platelets ≥100,000/mcL
   4. hemoglobin ≥ 9 g/dL (5.58 mmol/L)
   5. total bilirubin ≤1.5 x institutional upper limit of normal, unless attributed to Gilberts syndrome
   6. Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) < 2.5 x institutional upper limit of normal
   7. INR ≤1.5 x institutional upper limit of normal
   8. creatinine within normal institutional limits OR
   9. creatinine clearance ≥30 mL/min per Cockcroft-Gault formulation
   10. normal serum potassium, calcium, and magnesium levels (may be receiving supplements). Grade 1 hypocalcemia (corrected serum calcium > 8) is acceptable
10. Willing to undergo tumor biopsy prior to trial treatment, unless in the opinion of the treating physician, a biopsy is not feasible or safe. Subjects must be willing to ultimately undergo surgery if their tumor becomes surgically resectable
11. Ability to comply with outpatient treatment, laboratory monitoring, and require clinic visits for the duration of study participation
12. Willing and able to provide written informed consent signed by study patient (or legally acceptable representative if applicable)
13. Willingness of patients with partners of childbearing potential to use a highly effective contraceptive method during treatment with study drug and for 3 months following the last dose of study drug

Exclusion Criteria:

1. Radiographically identified following findings: intraluminal airway tumor, complete carotid encasement/infiltration
2. Patients with contraindications to the involved chemotherapy drugs (such as severe coagulopathy, severe liver function impairment, etc.)
3. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment
4. Gastrointestinal malabsorption or any other condition that in the opinion of the investigator might affect the absorption of study drug
5. Patients with serious internal medicine underlying diseases, serious organ dysfunction, metabolic diseases or other diseases that seriously affect survival
6. If > 1 + proteinuria on urine dipstick testing will undergo 24-hour urine collection for quantitative assessment of proteinuria. Participants with urine protein ≥1g/24 h will be ineligible
7. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction, or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment
8. Active hemoptysis (bright red blood ≥ 1/2 teaspoon) or other uncontrolled bleeding within 21 days prior to the study registration
9. Arterial/venous thromboembolic events in the last 12 months Treatment within 30 days prior to study registration with anticoagulant or antiplatelet therapy, apart from aspirin 81 mg daily
10. Active uncontrolled systemic bacterial, viral, or fungal infection, or serious ongoing intercurrent illness
11. Uncontrolled symptomatic hyperthyroidism or hypothyroidism
12. Females who are pregnant or breastfeeding
13. Other progressive malignant diseases requiring treatment
14. Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation, which must be completed at least 4 weeks prior to the first dose of study treatment
15. Symptomatic primary central nervous system (CNS) tumor, metastases, leptomeningeal carcinomatosis, or untreated spinal cord compression. Exception: Patients are eligible if neurological symptoms and CNS imaging are stable and no CNS surgery or radiation has been performed for 28 days, 14 days if stereotactic radiosurgery (SRS)
16. Patients with incomplete clinical data
17. History of significant neurological or mental disorder, including seizures or dementia, which would interfere compliance and sign of consent inform
18. Patients deemed unsuitable for inclusion by the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Every 2 months until 12 months
  To evaluate the efficacy of chemotherapy per RECIST (standard Response Evaluation Criteria in Solid Tumors [RECIST 1.1]), the percentages of patients will report that fall into each of the four categories: complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD)

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 2 years post treatment
  Defined as the time from patient registration to disease progression or death from any cause. Structural progression is defined according to RECIST criteria based on histopathologic findings, and biochemical progression is defined as abnormal thyroglobulin (Tg) or rising Tg antibody levels for anaplastic thyroid cancer/differentiated thyroid cancer, and abnormal carcinoembryonic antigen/calcitonin for medullary thyroid cancer
Overall survival (OS) | Up to 2 years post treatment
  Defined as the time from patient registration to death from any causes
R0/R1 resection rates | From the date of enrollment to the date of surgery, up to 12 months
  Defined by proportion of patients who undergo successful thyroidectomy with clear (R0) or microscopically positive (R1) surgical margins. Will evaluate R0/R1 resection rates in each of 4 pre-specified extrathyroidal anatomic target interfaces: 1) perithyroid muscles (e.g. strap, sternocleidomastoid, inferior constrictor muscles) 2) cartilage (larynx/trachea) 3) esophagus 4) recurrent laryngeal nerve
Incidence of adverse events | Every 2 months until 12 months
  Assessed as defined by Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0
Quality of life | Every 2 months until 12 months
  Assessed by the European Quality of Life 5 Dimension Questionnaire (EQ-5D). The EQ-5D consists of health state description and evaluation. The health state description consists of five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), with each dimension specifying five levels of severity [best (1)-worst (5)]. The health state evaluation is assessed using the visual analogue scale ([worse (0)-best (100)]

CONTACTS AND LOCATIONS:
Locations (1):
- West China hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No